CLINICAL TRIAL: NCT06351085
Title: Enhancing Lung Cancer Screening Through Human-Centered Intervention
Acronym: ELFE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Principal Investigator, Moon S. Chen,Jr. PhD,MPH, Principal Investigator, University of California, Davis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 1937769-1
Record Dates: First submitted 2024-03-26; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Lung Cancer
Keywords: Lung Cancer Screening
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: Patients of the intervention clinics will be assigned one of two interventions: 1) Pre Visit Planner (PVP) or 2) PVP + patient education delivered via the MyUCDHealth patient web portal.
Who Masked: Participant
Masking Description: Biostatistician created a randomized table to allocate patient in either intervention 1 or 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-Visit Planner (PVP) (Other): A Licensed Vocational Nurse (LVN) will verify patient smoking history and calculate pack years with the patient over the phone.
  Interventions: Behavioral: Pre-Visit Planner
- Pre-Visit Planner (PVP) + MyChart (Other): A Licensed Vocational Nurse (LVN) will verify patient smoking history and calculate pack years with the patient over the phone. In addition, the patient will receive educational video through MyChart prior to an LVN calling.
  Interventions: Behavioral: Pre-Visit Planner + MyChart
- Usual Care (No Intervention): Patients will receive usual care.

INTERVENTIONS:
Behavioral: Pre-Visit Planner — The study is comparing the implementation of a Pre-Visit Planner to go through the shared decision making process.
  Arms: Pre-Visit Planner (PVP)
Behavioral: Pre-Visit Planner + MyChart — The study is comparing the implementation of a Pre-Visit Planner to go through the shared decision making process as well as testing if watching educational videos about the Lung Cancer Screening (LCS) process prior to talking to an LVN will help with LCS uptake.
  Arms: Pre-Visit Planner (PVP) + MyChart

SUMMARY:
The purpose of this study is to further understand the factors involved in increasing lung cancer screening.

DETAILED DESCRIPTION:
The study aims to identify patient, primary care team and health system factors that facilitate participation in lung cancer screening. Additionally, conduct a two-arm randomized comparative effectiveness intervention study to increase lung cancer screening compared with a usual care control arm and further evaluate the differential impact of the intervention conditions compared to usual care.

ELIGIBILITY:
Inclusion Criteria:

Interviews:

* UC Davis Health Systems (UCDHS) primary care providers and clinic staff who provide services to patients ages 50-80.
* Patients who are eligible for lung cancer screening.

Screening Intervention:

- Patients ages 50-80 who have a history of smoking per review of their electronic medical record and who receive care at the following UCDH ambulatory care clinics: Ellison Ambulatory Care Clinic; Elk Grove; Midtown.

Exclusion Criteria:

Interviews:

* Non-consenting patients and patients who do not speak English or Spanish
* Patients aged 49 and younger
* Non UCDHS primary care providers and clinic staff

Screening Intervention:

* UCDHS patients who have already received Lung Cancer Screening
* Patients with existing Cancer diagnosis

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2869 (Estimated)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-04-14 (Estimated); Study Completion 2025-04-14 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Screening | 156 Weeks
  The primary outcome is the proportion of patients aged 50-80 with a history of smoking who receive Lung Cancer Screening during the study period; this outcome will be measured in both intervention groups and the control group.

SECONDARY OUTCOMES:
Completion of Interviews with Staff and Patients | 156 Weeks
  Key informant interviews with UC Davis staff and patients to determine approach to intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Davis, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No